CLINICAL TRIAL: NCT00289198
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study to Evaluate the Efficacy and Safety of Once-Daily Intranasal Administration of GW685698X Aqueous Nasal Spray 100mcg for 6 Weeks in Adult and Adolescent Subjects 12 Years of Age and Older With Perennial Allergic Rhinitis (PAR)
Brief Title: Once-Daily Investigational Nasal Spray In Adults And Adolescents With Perennial Allergic Rhinitis (PAR)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: FFR106080
Record Dates: First submitted 2006-02-08; First posted 2006-02-09 (Estimated); Results first posted 2018-04-13 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2017-09

CONDITIONS: Rhinitis, Allergic, Perennial
Keywords: GW685698X; perennial allergic rhinitis; allergic rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Rhinitis, Allergic

ARMS (2):
- Fluticasone furoate (Experimental): Participants were instructed to administer two sprays into each nostril once daily every morning of fluticasone furoate 110 μg
  Interventions: Drug: FF
- Placebo (Placebo Comparator): Participants were instructed to administer two sprays into each nostril once daily every morning of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FF — fluticasone furoate 110 μg nasal spray
  Arms: Fluticasone furoate
Drug: Placebo — placebo nasal spray
  Arms: Placebo

SUMMARY:
The primary objective of this study is to compare the efficacy and safety of GW685698X 100mcg once daily (QD) aqueous nasal spray with vehicle placebo nasal spray in adult and adolescent subjects (12 years of age and older) with perennial allergic rhinitis (PAR).

DETAILED DESCRIPTION:
A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study to Evaluate the Efficacy and Safety of Once-Daily Intranasal Administration of GW685698X Aqueous Nasal Spray 100mcg for 6 Weeks in Adult and Adolescent Subjects 12 years of Age and Older with Perennial Allergic Rhinitis (PAR)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of perennial allergic rhinitis (PAR).
* Must comply with study procedures and be literate.

Exclusion Criteria:

* Significant concomitant medical conditions.
* Use of corticosteroids.
* Use of allergy and other identified medications during the study.
* Current tobacco use or tobacco use within the past year.
* Exposure to an investigational study drug within the past 12 months.
* Clinically significant abnormal electrocardiograms (ECG) or laboratory abnormality.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2006-02-07; Primary Completion 2006-07-01 (Actual); Study Completion 2006-07-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (35):
- United States (8):
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Wheaton, Maryland
  - GSK Investigational Site, North Dartmouth, Massachusetts
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, South Burlington, Vermont
- Australia (7):
  - GSK Investigational Site, Camperdown, New South Wales
  - GSK Investigational Site, Kippa-Ring, Queensland
  - GSK Investigational Site, Toorak Gardens, South Australia
  - GSK Investigational Site, Clayton, Victoria
  - GSK Investigational Site, Melbourne, Victoria
  - GSK Investigational Site, Parkville, Victoria
  - GSK Investigational Site, Nedlands, Western Australia
- Canada (4):
  - GSK Investigational Site, Mississauga, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Trois-Rivières, Quebec
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Germany (3):
  - GSK Investigational Site, Schwerin, Mecklenburg-Vorpommern
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Latvia (4):
  - GSK Investigational Site, Dobele
  - GSK Investigational Site, Liepāja
  - GSK Investigational Site, Riga
  - GSK Investigational Site, Tukums
- Lithuania (3):
  - GSK Investigational Site, Kaunas
  - GSK Investigational Site, Šiauliai
  - GSK Investigational Site, Vilnius
- New Zealand (2):
  - GSK Investigational Site, Auckland
  - GSK Investigational Site, Grafton
- Russia (2):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: FFR106080 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: FFR106080 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: FFR106080 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: FFR106080 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: FFR106080 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: FFR106080 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: FFR106080 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from 07 February 2006 till 23 June 2006 at 40 centers across the globe. A total of 288 participants with perennial allergic rhinitis (PAR) were planned to be enrolled.
Pre-assignment Details: Following a 7 to 14 day screening period, participants who met randomisation criteria were randomised to 6 weeks of treatment with fluticasone furoate or placebo nasal spray once daily. A total of 302 participants were randomised, 151 in each of the treatment groups.
Groups:
- Placebo: Eligible participants received aqueous nasal spray of matching Placebo once daily for 6 weeks in a randomized manner. Dose was administered by alternately spraying one spray into each nostril followed by a second spray into each nostril for 42 days. Participants were followed-up telephonically, up to 5 days after the last dose of the study drug.
- Fluticasone Furoate: Eligible participants received aqueous nasal spray of Fluticasone furoate 100 micrograms (mcg) once daily for 6 weeks in a randomized manner. Dose was administered by alternately spraying one spray (27.5 mcg per spray) into each nostril followed by a second spray into each nostril for 42 days. Participants were followed-up telephonically, up to 5 days after the last dose of the study drug.
Period: Overall Study
Arm/Group | Placebo | Fluticasone Furoate
Started | 151 | 151
Completed | 120 | 121
Not Completed | 31 | 30
Not completed — Adverse Event | 0 | 2
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Lack of Efficacy | 2 | 0
Not completed — Other: Low compliance | 0 | 1
Not completed — Other: Physician's decision | 0 | 1
Not completed — Other: Unable to attend on schedule | 2 | 1
Not completed — Other: Miscalculation of the visit date | 21 | 22
Not completed — Other: Impossible to come on visit | 0 | 1

BASELINE CHARACTERISTICS:
Population: The ITT Population included all participants who were randomized and received at least one dose of the study drug.
Groups:
- Fluticasone Furoate: Eligible participants received aqueous nasal spray of Fluticasone furoate 100 mcg once daily for 6 weeks in a randomized manner. Dose was administered by alternately spraying one spray into each nostril followed by a second spray into each nostril for 42 days. Participants were followed-up telephonically, up to 5 days after the last dose of the study drug.
- Total: Total of all reporting groups
Arm/Group | Fluticasone Furoate | Placebo | Total
Number analyzed (Participants) | 151 | 151 | 302
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.1 (16.57) | 37.2 (16.20) | 37.1 (16.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 86 | 171
  Male | 66 | 65 | 131
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 4 | 3 | 7
  American Indian or Alaska Native | 0 | 1 | 1
  Asian - Central/South Asian Heritage | 2 | 1 | 3
  Asian - East Asian Heritage | 1 | 1 | 2
  Asian - South East Asian Heritage | 6 | 4 | 10
  Native Hawaiian or other Pacific Islander | 3 | 0 | 3
  White - Arabic/North African Heritage | 0 | 1 | 1
  White - White/Caucasian/European Heritage | 135 | 139 | 274
  Mixed Race | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline (Day 1) Over the Entire Treatment Period in Daily, Reflective Total Nasal Symptom Scores (rTNSS) Over 6 Weeks
Description: TNSS is the sum of symptom scores for rhinorrhea, nasal congestion, nasal itching, and sneezing (each scored on a scale of 0 [none] to 3 [severe]; total possible score of 0 to 12). The rTNSS is a rating of the severity of symptoms over the previous 12 hours and is performed in morning (AM) and evening (PM). Daily rTNSS is defined as average of the PM rTNSS and the AM rTNSS of the next day prior to AM dosing. The Baseline daily rTNSS is defined as the average of the daily rTNSS over 4 consecutive 24 hour periods prior to randomization plus randomization day AM assessment. Change from Baseline was calculated as average of the non-missing daily rTNSS minus Baseline daily rTNSS. Analysis was performed using analysis of covariance (ANCOVA), adjusting for Baseline daily rTNSS, country, age, and gender. The Intent To Treat (ITT) Population comprised of all randomized participants who received >=1 dose of study drug. Only those participants available at the specified time points were analyzed
Time Frame: Baseline (Day 1) and up to Week 6
Population: ITT population. Data is presented for the participants available at the time of assessment.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Fluticasone Furoate
Number analyzed (Participants) | 150 | 151
Scores on a scale | -2.69 (0.18) | -3.95 (0.18)
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Furoate; Test type: Superiority or Other; p < 0.001, ANCOVA — Change from Baseline (Day 1) in reflective total nasal symptom scores for Placebo versus that for fluticasone furoate; Mean Difference (Final Values) = -1.256, 95% CI 2-sided [-1.73 to -0.78]

2. Secondary Outcome: Mean Change From Baseline (Day 1) in AM, Pre-dose, Instantaneous Total Nasal Symptom (iTNSS) Scores Over the Entire Treatment Period
Description: The AM pre-dose iTNSS is the sum of the 4 individual nasal symptom score assessments for rhinorrhea, nasal congestion, nasal itching, and sneezing performed at the moment immediately prior to taking the daily dose; each individual symptom score ranged on a scale of 0 to 3 where 0 indicated healthy condition and 3 indicated severity of the symptoms. The total score ranged on a scale of 0 to 12 where 0 indicated healthy condition and 12 indicated worst condition of symptoms. Baseline iTNSS is defined as the average of the non-missing values for iTNSS during the Baseline period where the Baseline period included the randomization day and the 3 consecutive days prior to randomization. Change from Baseline was calculated as score over the entire treatment period minus Baseline value. Analysis was performed using ANCOVA, adjusting for Baseline value, country, age, and gender. Only those participants available at the specified time points were analyzed.
Time Frame: Baseline (Day 1) and up to Week 6
Population: ITT population. Data is presented for the participants available at the time of assessment.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Fluticasone Furoate
Number analyzed (Participants) | 149 | 150
Scores on a scale | -2.36 (0.18) | -3.82 (0.18)
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Furoate; Test type: Superiority or Other; p < 0.001, ANCOVA — Mean change from Baseline in AM pre-dose instantaneous TNSS over entire period for Placebo versus that for Fluticasone furoate; Mean Difference (Final Values) = -1.459, 95% CI 2-sided [-1.93 to -0.99]

3. Secondary Outcome: Number of Participants With Response to Therapy Over Entire Treatment Period
Description: Response to therapy is defined as the effectiveness of FF for relieving allergic rhinitis symptoms over the entire treatment period. Response was, evaluated at the end of the study (Week 6) using a 7-point categorical scale, categorized as: 1=significantly improved, 2=moderately improved, 3=mildly improved, 4=no change, 5=mildly worse, 6=moderately worse, 7=significantly worse. Analysis was performed using logistic regression to evaluate treatment effect, adjusting for age, gender, and country. Effectiveness of the study drug for relieving allergic rhinitis symptoms over the entire treatment period was compared with Placebo.
Time Frame: Up to 6 weeks
Population: ITT population. Data is presented for the participants available at the time of assessment.
Measure: Number; unit: Participants
Arm/Group | Placebo | Fluticasone Furoate
Number analyzed (Participants) | 151 | 151
Participants
  Significantly Improved | 21 | 56
  Moderately Improved | 38 | 37
  Mildly Improved | 37 | 31
  No Change | 45 | 20
  Mildly Worse | 5 | 2
  Moderately Worse | 3 | 3
  Significantly Worse | 2 | 2
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Furoate; Test type: Superiority; p < 0.001, Regression, Logistic; Based on logistic regression adjusting for age, gender and country

4. Secondary Outcome: Mean Change From Baseline (Day 1) in AM rTNSS Over the Entire Treatment Period
Description: TNSS is the sum of symptom scores for rhinorrhea, nasal congestion, nasal itching, and sneezing (each scored on a scale of 0 [none] to 3 [severe]; total possible score of 0 to 12). The AM rTNSS is a rating of the severity of symptoms performed in the morning prior to administering the dose of study drug and assesses how the participant felt during the night (preceding 12 hours). Baseline rTNSS is defined as the average of the non-missing values for rTNSS during the Baseline period where the Baseline period included the randomization day and the 3 consecutive days prior to randomization. Change from Baseline was calculated as score over the entire treatment period minus Baseline value. Analysis was performed using ANCOVA, adjusting for Baseline value, country, age, and gender. Only those participants available at the specified time points were analyzed.
Time Frame: Baseline (Day 1) and up to 6 weeks
Population: ITT population. Data is presented for the participants available at the time of assessment.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Fluticasone Furoate
Number analyzed (Participants) | 149 | 150
Scores on a scale | -2.66 (0.17) | -3.93 (0.17)
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Furoate; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -1.274, 95% CI 2-sided [-1.74 to -0.81]

5. Secondary Outcome: Mean Change From Baseline (Day 1) in PM rTNSS Over the Entire Treatment Period
Description: TNSS is the sum of symptom scores for rhinorrhea, nasal congestion, nasal itching, and sneezing (each scored on a scale of 0 [none] to 3 [severe]; total possible score of 0 to 12). The PM rTNSS is a rating of the severity of symptoms performed approximately 12 hours after dosing and before bedtime and assesses how the participant felt during the day. Baseline rTNSS is defined as the average of the non-missing values for rTNSS during the Baseline period where the baseline period includes the 4 consecutive days prior to randomization. Change from Baseline was calculated as score over the entire treatment period minus Baseline value. Analysis was performed using ANCOVA, adjusting for Baseline value, country, age, and gender. Only those participants available at the specified time points were analyzed.
Time Frame: Baseline (Day 1) and up to 6 weeks
Population: ITT population. Data is presented for the participants available at the time of assessment.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Fluticasone Furoate
Number analyzed (Participants) | 150 | 150
Scores on a scale | -2.73 (0.18) | -4.02 (0.18)
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Furoate; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -1.291, 95% CI 2-sided [-1.77 to -0.81]

6. Secondary Outcome: Mean Percent Change From Baseline (Day 1) in Daily rTNSS Over the Entire Treatment Period
Description: as for outcome 1
Time Frame: Baseline (Day 1) and up to 6 weeks
Population: ITT population. Data is presented for the participants available at the time of assessment.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Fluticasone Furoate
Number analyzed (Participants) | 150 | 151
Percent change | -30.23 (2.22) | -44.35 (2.21)
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Furoate; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -14.118, 95% CI 2-sided [-20.03 to -8.21]

7. Secondary Outcome: Mean Percent Change From Baseline (Day 1) in AM Pre-Dose iTNSS Over the Entire Treatment Period
Description: TNSS is the sum of symptom scores for rhinorrhea, nasal congestion, nasal itching, and sneezing (each scored on a scale of 0 [none] to 3 [severe]; total possible score of 0 to 12). The rTNSS is a rating of the severity of symptoms over the previous 12 hours and is performed in morning (AM) and evening (PM). Daily rTNSS is defined as average of the PM rTNSS and the AM rTNSS of the next day prior to AM dosing. The BL daily rTNSS is defined as the average of the daily rTNSS over 4 consecutive 24-hour periods prior to randomization plus randomization day AM assessment. Change from Baseline was calculated as average of the non-missing daily rTNSS minus Baseline daily rTNSS. Analysis was performed using ANCOVA, adjusting for BL daily rTNSS, country, age, and gender. Only those participants available at the specified time points were analyzed. Change from Baseline is the value at indicated time-point minus the baseline value*100.
Time Frame: Baseline and up to 6 weeks
Population: ITT population. Data is presented for the participants available at the time of assessment.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Fluticasone Furoate
Number analyzed (Participants) | 149 | 150
Percent change | -24.67 (2.66) | -44.70 (2.66)
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Furoate; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -20.033, 95% CI 2-sided [-27.13 to -12.94]

8. Secondary Outcome: Mean Change From Baseline (Day 1) in Daily Reflective Individual Nasal Symptom Scores (rINSS) Over the Entire Treatment Period
Description: The individual nasal symptom scores (INSS) for rhinorrhea, nasal congestion, nasal itching and sneezing were assessed on a 4 point (0 [none] to 3 [severe]) categorical scale and larger score indicates severe symptoms. The INSS is a rating of the severity of symptoms over the previous 12 hours and is performed in AM and PM. Daily INSS is defined as average of the PM INSS and the AM INSS of the next day prior to AM dosing. The Baseline daily INSS is defined as the average of the daily INSS over 4 consecutive 24-hour periods prior to randomization plus randomization day AM assessment. Change from Baseline was calculated as average of the non-missing daily INSS minus Baseline daily INSS. Analysis was performed using ANCOVA, adjusting for Baseline value, country, age, and gender.
Time Frame: Baseline (Day 1) and up to 6 weeks
Population: ITT population. Only those participants available at the time of assessment were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Fluticasone Furoate
Number analyzed (Participants) | 150 | 151
Scores on a scale
  Rhinorrhea | -0.67 (0.05) | -0.94 (0.05)
  Nasal Congestion | -0.69 (0.05) | -0.97 (0.05)
  Nasal Itching | -0.65 (0.05) | -0.98 (0.05)
  Sneezing | -0.68 (0.05) | -1.07 (0.05)
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Furoate; Rhinorrhea score, Placebo vs Fluticasone furoate; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -0.277, 95% CI 2-sided [-0.41 to -0.14]
Statistical Analysis 2: Comparison: Placebo vs Fluticasone Furoate; Nasal Congestion, Placebo vs Fluticasone furoate; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -0.277, 95% CI 2-sided [-0.42 to -0.14]
Statistical Analysis 3: Comparison: Placebo vs Fluticasone Furoate; Nasal Itching, Placebo vs Fluticasone furoate; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -0.331, 95% CI 2-sided [-0.47 to -0.20]
Statistical Analysis 4: Comparison: Placebo vs Fluticasone Furoate; Sneezing score, Placebo vs Fluticasone furoate; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -0.390, 95% CI 2-sided [-0.52 to -0.27]

9. Secondary Outcome: Mean Change From Baseline (Day 1) in AM Pre-dose Instantaneous Individual Nasal Symptom Score (iINSS) Over the Entire Treatment Period
Description: The iINSS score for rhinorrhea, nasal congestion, nasal itching and sneezing were assessed on a 4 point (0 [none] to 3 [severe]) categorical scale and larger score indicates severe symptoms. The AM pre-dose iINSS is a rating of the severity of symptoms performed at the moment immediately prior to dosing. Baseline iINSS is defined as the average of the non-missing values for iINSS during the Baseline period where the Baseline period included the randomization day and the 3 consecutive days prior to randomization. Change from Baseline was calculated as score over the entire treatment period minus Baseline value. Analysis was performed using ANCOVA, adjusting for Baseline value, country, age, and gender. Only those participants available at the specified time points were analyzed.
Time Frame: Baseline (Day 1) and up to 6 weeks
Population: ITT population. Data is presented for the participants available at the time of assessment.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Fluticasone Furoate
Number analyzed (Participants) | 149 | 150
Scores on a scale
  Rhinorrhea | -0.57 (0.05) | -0.93 (0.05)
  Nasal Congestion | -0.55 (0.05) | -0.92 (0.05)
  Nasal Itching | -0.61 (0.05) | -0.98 (0.05)
  Sneezing | -0.63 (0.05) | -1.00 (0.05)
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Furoate; Rhinorrhea score, Placebo versus fluticasone furoate; Test type: Superiority or Other; p = 0.001, ANCOVA; Mean Difference (Final Values) = -0.357, 95% CI 2-sided [-0.50 to -0.22]
Statistical Analysis 2: Comparison: Placebo vs Fluticasone Furoate; Nasal Congestion score, Placebo versus fluticasone furoate; Test type: Superiority or Other; p = 0.001, ANCOVA; Mean Difference (Final Values) = -0.370, 95% CI 2-sided [-0.51 to -0.23]
Statistical Analysis 3: Comparison: Placebo vs Fluticasone Furoate; Nasal itching score, Placebo versus fluticasone furoate; Test type: Superiority or Other; p = 0.001, ANCOVA; Mean Difference (Final Values) = -0.372, 95% CI 2-sided [-0.50 to -0.24]
Statistical Analysis 4: Comparison: Placebo vs Fluticasone Furoate; Sneezing score, Placebo versus fluticasone furoate; Test type: Superiority or Other; p = 0.001, ANCOVA; Mean Difference (Final Values) = -0.372, 95% CI 2-sided [-0.50 to -0.24]

10. Secondary Outcome: Mean Change From Baseline (Day 1) in AM rINSS Over the Entire Treatment
Description: INSS for rhinorrhea, nasal congestion, nasal itching and sneezing were assessed on a 4 point (0 [none] to 3 [severe]) categorical scale and larger score indicates severe symptoms. The AM rINSS is a rating of the severity of symptoms performed in the morning prior to administering the dose of study drug and assesses how the participant felt during the night (preceding 12 hours). Baseline rINSS is defined as the average of the non-missing values for rINSS during the Baseline period where the Baseline period included the randomization day and the 3 consecutive days prior to randomization. Change from Baseline was calculated as score over the entire treatment period minus Baseline value. Analysis was performed using ANCOVA, adjusting for Baseline value, country, age, and gender. Only those par. available at the specified time points were analyzed.
Time Frame: Baseline (Day 1) and up to 6 weeks
Population: ITT population. Data is presented for the participants available at the time of assessment.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Fluticasone Furoate
Number analyzed (Participants) | 149 | 150
Scores on a scale
  Rhinorrhea | -0.67 (0.05) | -0.95 (0.05)
  Nasal Congestion | -0.66 (0.05) | -0.98 (0.05)
  Nasal Itching | -0.64 (0.05) | -0.96 (0.05)
  Sneezing | -0.69 (0.05) | -1.06 (0.05)
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Furoate; Rhinorrhea score,Placebo versus fluticasone furoate; Test type: Superiority or Other; p = 0.001, ANCOVA; Mean Difference (Final Values) = -0.281, 95% CI 2-sided [-0.42 to -0.14]
Statistical Analysis 2: Comparison: Placebo vs Fluticasone Furoate; Nasal Congestion score, Placebo versus fluticasone furoate; Test type: Superiority or Other; p = 0.001, ANCOVA; Mean Difference (Final Values) = -0.314, 95% CI 2-sided [-0.45 to -0.17]
Statistical Analysis 3: Comparison: Placebo vs Fluticasone Furoate; Nasal itching score, Placebo versus fluticasone furoate; Test type: Superiority or Other; p = 0.001, ANCOVA; Mean Difference (Final Values) = -0.324, 95% CI 2-sided [-0.45 to -0.19]
Statistical Analysis 4: Comparison: Placebo vs Fluticasone Furoate; Sneezing score, Placebo versus fluticasone furoate; Test type: Superiority or Other; p = 0.001, ANCOVA; Mean Difference (Final Values) = -0.374, 95% CI 2-sided [-0.50 to -0.25]

11. Secondary Outcome: Mean Change From Baseline (Day 1) in PM rINSS Over the Entire Treatment Period
Description: rINSS for rhinorrhea, nasal congestion, nasal itching and sneezing were assessed on a 4 point (0 [none] to 3 [severe]) categorical scale and larger score indicates severe symptoms. The PM rINSS is a rating of the severity of symptoms performed approximately 12 hours after dosing and before bedtime and assesses how the participant felt during the day. Baseline rINSS is defined as the average of the non-missing values for rINSS during the Baseline period where the Baseline period included the 4 consecutive days prior to randomization. Change from Baseline was calculated as score over the entire treatment period minus Baseline value. Analysis was performed using ANCOVA, adjusting for Baseline value, country, age, and gender. Only those par. available at the specified time points were analyzed.
Time Frame: Baseline (Day 1) and up to 6 weeks
Population: ITT population
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Groups:
- Fluticasone Furoate: Eligible participants received aqueous nasal spray of Fluticasone furoate 100 micrograms (mcg) once daily for 6 weeks in a randomized manner. Dose was administered by alternately spraying one spray into each nostril followed by a second spray into each nostril for 42 days. Participants were followed-up telephonically, up to 5 days after the last dose of the study drug.
Arm/Group | Placebo | Fluticasone Furoate
Number analyzed (Participants) | 150 | 150
Scores on a scale
  Rhinorrhea | -0.66 (0.05) | -0.96 (0.05)
  Nasal Congestion | -0.70 (0.05) | -0.97 (0.05)
  Nasal Itching | -0.68 (0.05) | -1.01 (0.05)
  Sneezing | -0.68 (0.05) | -1.09 (0.05)
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Furoate; Rhinorrhea score, Placebo vs Fluticasone furoate; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -0.292, 95% CI [-0.43 to -0.15]
Statistical Analysis 2: Comparison: Placebo vs Fluticasone Furoate; Nasal Congestion score, Placebo vs Fluticasone furoate; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -0.264, 95% CI 2-sided [-0.40 to -0.12]
Statistical Analysis 3: Comparison: Placebo vs Fluticasone Furoate; Nasal Itching score, Placebo vs Fluticasone furoate; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -0.336, 95% CI 2-sided [-0.48 to -0.20]
Statistical Analysis 4: Comparison: Placebo vs Fluticasone Furoate; Sneezing score, Placebo vs Fluticasone furoate; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -0.412, 95% CI 2-sided [-0.54 to -0.28]

12. Secondary Outcome: Mean Change From Baseline (Day 1) in Daily Reflective Total Ocular Symptom Score (rTOSS) Over the Entire Treatment Period
Description: TOSS is defined as the sum of the 3 individual ocular symptom scores for itching/burning eyes, tearing/watering eyes, and eye redness, and ranges from 0 to 9. Each symptom is scored on a 4 point (0 [none] to 3 [severe]) categorical scale. The rTOSS is a rating of the severity of symptoms over the previous 12 hours and is performed in AM and PM. Daily rTOSS is defined as average of the PM rTOSS and the AM rTOSS of the next day prior to AM dosing. The BL daily rTOSS is defined as the average of the daily rTOSS over 4 consecutive 24-hour periods prior to randomization plus randomization day AM assessment. Change from BL was calculated as average of the non-missing daily rTOSS minus BL daily rTOSS. Analysis was performed using ANCOVA, adjusting for BL value, country, age, and gender. Only those participants available at the specified time points were analyzed.
Time Frame: Baseline (Day 1) and up to 6 weeks
Population: ITT population. Data is presented for the participants available at the time of assessment.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Fluticasone Furoate
Number analyzed (Participants) | 150 | 151
Scores on a scale | -1.41 (0.13) | -1.92 (0.13)
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Furoate; Test type: Superiority or Other; p = 0.004, ANCOVA; Mean Difference (Final Values) = -0.506, 95% CI 2-sided [-0.85 to -0.16]

13. Secondary Outcome: Mean Change From Baseline (Day 1) in AM Pre-dose Instantaneous TOSS (iTOSS) Over the Entire Treatment Period
Description: The TOSS score is defined as the sum of the 3 individual ocular symptom scores for itching/burning eyes, tearing/watering eyes, and eye redness, and ranges from 0 to 9. Each symptom is scored on a 4 point (0 [none] to 3 [severe]) categorical scale. The AM pre-dose iTOSS is a rating of the severity of symptoms performed at the moment immediately prior to dosing. Baseline iTOSS is defined as the average of the non-missing values for iTOSS during the Baseline period where the Baseline period included the randomization day and the 3 consecutive days prior to randomization. Change from Baseline was calculated as score over the entire treatment period minus Baseline value. Analysis was performed using ANCOVA, adjusting for Baseline value, country, age, and gender.
Time Frame: Baseline (Day 1) and up to 6 weeks
Population: ITT population. Data is presented for the participants available at the time of assessment.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Fluticasone Furoate
Number analyzed (Participants) | 149 | 150
Scores on a scale | -1.26 (0.13) | -1.76 (0.13)
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Furoate; Test type: Superiority or Other; p = 0.007, ANCOVA; Mean Difference (Final Values) = -0.491, 95% CI [-0.85 to -0.13]

14. Secondary Outcome: Mean Change From Baseline (Day 1) in AM rTOSS Over the Entire Treatment Period
Description: The TOSS score is defined as the sum of the 3 individual ocular symptom scores for itching/burning eyes, tearing/watering eyes, and eye redness, and ranges from 0 to 9. Each symptom is scored on a 4 point (0 [none] to 3 [severe]) categorical scale and larger score indicates more severe symptoms. The AM rTOSS is a rating of the severity of symptoms performed in the morning prior to administering the dose of study drug and assesses how the participant felt during the night (preceding 12 hours). Baseline rTOSS is defined as the average of the non-missing values for rTOSS during the Baseline period where the Baseline period includes the randomization day and the 3 consecutive days prior to randomization. Change from Baseline was calculated as score over the entire treatment period minus Baseline value. Analysis was performed using ANCOVA, adjusting for Baseline value, country, age, and gender. Only those participants available at the specified time points were analyzed
Time Frame: Baseline (Day 1) and up to 6 weeks
Population: ITT population. Data is presented for the participants available at the time of assessment.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Fluticasone Furoate
Number analyzed (Participants) | 149 | 150
Scores on a scale | -1.39 (0.13) | -1.92 (0.13)
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Furoate; Test type: Superiority or Other; p = 0.003, ANCOVA; Mean Difference (Final Values) = -0.531, 95% CI 2-sided [-0.88 to -0.19]

15. Secondary Outcome: Mean Change From Baseline (Day 1) in PM rTOSS Over the Entire Treatment Period
Description: The TOSS score is defined as the sum of the 3 individual ocular symptom scores for itching/burning eyes, tearing/watering eyes, and eye redness, and ranges from 0 to 9. Each symptom is scored on a 4 point (0 [none] to 3 [severe]) categorical scale. The PM rTOSS is a rating of the severity of symptoms performed approximately 12 hours after dosing and before bedtime and assesses how the participant felt during the day. Baseline rTOSS is defined as the average of the non-missing values for rTOSS during the Baseline period where the baseline period includes the 4 consecutive days prior to randomization. Change from Baseline was calculated as score over the entire treatment period minus Baseline value. Analysis was performed using ANCOVA, adjusting for Baseline value, country, age, and gender. Only those participants available at the specified time points were analyzed.
Time Frame: Baseline (Day 1) and up to 6 weeks
Population: ITT population. Data is presented for the participants available at the time of assessment.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Fluticasone Furoate
Number analyzed (Participants) | 150 | 150
Scores on a scale | -1.44 (0.13) | -1.93 (0.13)
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Furoate; Test type: Superiority or Other; p = 0.005, ANCOVA; Mean Difference (Final Values) = -0.496, 95% CI 2-sided [-0.84 to -0.15]

16. Secondary Outcome: Mean Change From Baseline (Day 1) in Daily Reflective Individual Ocular Symptom Scores (iIOSS) Over the Entire Treatment Period
Description: Individual ocular symptom scores (IOSS) for itching/burning eyes, tearing/watering eyes, and eye redness were assessed on a 4 point (0 [none]to 3 [severe]) categorical scale. The IOSS is a rating of the severity of symptoms over the previous 12 hours and is performed in AM and PM. Daily IOSS is defined as average of the PM IOSS and the AM IOSS of the next day prior to AM dosing. The BL daily IOSS is defined as the average of the daily IOSS over 4 consecutive 24-hour periods prior to randomization plus randomization day AM assessment. Change from BL was calculated as average of the non-missing daily IOSS minus BL daily IOSS. Analysis was performed using ANCOVA, adjusting for BL value, country, age, and gender.
Time Frame: Baseline (Day 1) and up to 6 weeks
Population: ITT population. Data is presented for the participants available at the time of assessment.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Fluticasone Furoate
Number analyzed (Participants) | 150 | 151
Scores on a scale
  Eye itching/burning | -0.47 (0.05) | -0.69 (0.05)
  Eye tearing/watering | -0.48 (0.05) | -0.62 (0.05)
  Eye redness | -0.45 (0.04) | -0.61 (0.04)
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Furoate; Eye itching/burning score, Placebo vs fluticasone furoate; Test type: Superiority or Other; p = 0.001, ANCOVA; Mean Difference (Final Values) = -0.216, 95% CI 2-sided [-0.34 to -0.09]
Statistical Analysis 2: Comparison: Placebo vs Fluticasone Furoate; Eye tearing/watering score, Placebo vs fluticasone furoate; Test type: Superiority or Other; p = 0.028, ANCOVA; Mean Difference (Final Values) = -0.137, 95% CI 2-sided [-0.26 to -0.02]
Statistical Analysis 3: Comparison: Placebo vs Fluticasone Furoate; Eye redness, Placebo vs fluticasone furoate; Test type: Superiority or Other; p = 0.010, ANCOVA; Mean Difference (Final Values) = -0.156, 95% CI 2-sided [-0.27 to -0.04]

17. Secondary Outcome: Mean Change From Baseline (Day 1) in AM Pre-Dose Instantaneous Individual Ocular Symptom Score (iIOSS) Over the Entire Treatment Period
Description: IOSS for itching/burning eyes, tearing/watering eyes, and eye redness were assessed on a 4 point (0 [none]to 3 [severe]) categorical scale. The AM pre-dose iIOSS is a rating of the severity of symptoms performed at the moment immediately prior to dosing. Baseline iIOSS is defined as the average of the non-missing values for iIOSS during the Baseline period where the Baseline period includes the randomization day and the 3 consecutive days prior to randomization. Change from Baseline is calculated as the score over the entire treatment period minus the score at Baseline. Analysis was performed using ANCOVA, adjusting for Baseline value, country, age, and gender.
Time Frame: Baseline (Day 1) and up to 6 weeks
Population: ITT population. Data is presented for the participants available at the time of assessment.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Fluticasone Furoate
Number analyzed (Participants) | 149 | 150
Scores on a scale
  Eye itching/burning | -0.39 (0.05) | -0.6 (0.5)
  Eye tearing/watering | -0.43 (0.05) | -0.59 (0.05)
  Eye redness | -0.45 (0.05) | -0.56 (0.05)
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Furoate; Eye itching/burning score, Placebo vs fluticasone furoate; Test type: Superiority or Other; p = 0.002, ANCOVA; Mean Difference (Final Values) = -0.215, 95% CI 2-sided [-0.35 to -0.08]
Statistical Analysis 2: Comparison: Placebo vs Fluticasone Furoate; Eye tearing or watering, Placebo vs fluticasone furoate; Test type: Superiority or Other; p = 0.016, ANCOVA; Mean Difference (Final Values) = -0.161, 95% CI [-0.29 to -0.03]
Statistical Analysis 3: Comparison: Placebo vs Fluticasone Furoate; Eye redness score, Placebo vs fluticasone furoate; Test type: Superiority or Other; p = 0.076, ANCOVA; Mean Difference (Final Values) = -0.113, 95% CI 2-sided [-0.24 to -0.01]

18. Secondary Outcome: Mean Change From Baseline (Day 1) in AM Reflective Individual Ocular Symptom Score (rIOSS) Over the Entire Treatment Period
Description: rIOSS for itching/burning eyes, tearing/watering eyes, and eye redness were assessed on a 4 point (0 [none]to 3 [severe]) categorical scale. The AM rIOSS is a rating of the severity of symptoms performed in the morning prior to administering the dose of study drug and assesses how the participant felt during the night (preceding 12 hours). Baseline rIOSS is defined as the average of the non-missing values for rIOSS during the Baseline period where the Baseline period includes the randomization day and the 3 consecutive days prior to randomization. Change from Baseline was calculated as score over the entire treatment period minus Baseline value. Analysis was performed using ANCOVA, adjusting for Baseline value, country, age, and gender.
Time Frame: Baseline (Day 1) and up to 6 weeks
Population: ITT population. Data is presented for the participants available at the time of assessment.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Fluticasone Furoate
Number analyzed (Participants) | 149 | 150
Scores on a scale
  Eye itching/burning | -0.48 (0.05) | -0.69 (0.05)
  Eye tearing/watering | -0.48 (0.05) | -0.62 (0.05)
  Eye redness | -0.44 (0.05) | -0.61 (0.05)
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Furoate; Eye itching/burning score, Placebo vs Fluticasone furoate; Test type: Superiority or Other; p = 0.001, ANCOVA; Mean Difference (Final Values) = -0.211, 95% CI 2-sided [-0.34 to -0.08]
Statistical Analysis 2: Comparison: Placebo vs Fluticasone Furoate; Eye tearing/watering, Placebo vs Fluticasone furoate; Test type: Superiority or Other; p = 0.023, ANCOVA; Mean Difference (Final Values) = -0.145, 95% CI 2-sided [-0.27 to -0.02]
Statistical Analysis 3: Comparison: Placebo vs Fluticasone Furoate; Eye Redness score, Placebo vs Fluticasone furoate; Test type: Superiority or Other; p = 0.005, ANCOVA; Mean Difference (Final Values) = -0.176, 95% CI 2-sided [-0.30 to -0.05]

19. Secondary Outcome: Mean Change From Baseline (Day 1) in PM rIOSS Over the Entire Treatment Period
Description: IOSS for itching/burning eyes, tearing/watering eyes, and eye redness were assessed on a 4 point (0 [none]to 3 [severe]) categorical scale. The PM rIOSS is a rating of the severity of symptoms performed approximately 12 hours after dosing and before bedtime and assesses how the participant felt during the day. Baseline rIOSS is defined as the average of the non-missing values for rIOSS during the Baseline period where the baseline period includes the 4 consecutive days prior to randomization. Change from Baseline is calculated as the score over the entire treatment period minus the score at Baseline. Analysis was performed using ANCOVA, adjusting for Baseline value, country, age, and gender.
Time Frame: Baseline (Day 1) and up to 6 weeks
Population: ITT population. Data is presented for the participants available at the time of assessment.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Fluticasone Furoate
Number analyzed (Participants) | 150 | 150
Scores on a scale
  Eye itching/burning | -0.47 (0.05) | -0.69 (0.05)
  Eye tearing/watering | -0.49 (0.05) | -0.62 (0.05)
  Eye redness | -0.47 (0.05) | -0.61 (0.05)
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Furoate; Eye itching/burning, Placebo vs fluticasone furoate; Test type: Superiority or Other; p = 0.001, ANCOVA; Mean Difference (Final Values) = -0.223, 95% CI 2-sided [-0.35 to -0.09]
Statistical Analysis 2: Comparison: Placebo vs Fluticasone Furoate; Eye Tearing/Watering score, Placebo vs fluticasone furoate; Test type: Superiority or Other; p = 0.040, ANCOVA; Mean Difference (Final Values) = -0.130, 95% CI 2-sided [-0.25 to -0.01]
Statistical Analysis 3: Comparison: Placebo vs Fluticasone Furoate; Eye Redness score, Placebo vs fluticasone furoate; Test type: Superiority or Other; p = 0.022, ANCOVA; Mean Difference (Final Values) = -0.142, 95% CI 2-sided [-0.26 to -0.02]

20. Secondary Outcome: Mean Change From Baseline (Day 1) in Daily Peak Nasal Inspiratory Flow (PNIF) Over the Entire Treatment Period
Description: PNIF is the tool for determining the extent of nasal airway obstruction. Participants used a portable hand-held inspiratory flow meter and face mask to measure and record PNIF. PNIF measurements was completed and recorded following assessment of allergy symptoms in the AM (prior to taking study medication), and 12 hours later in the PM (after recording allergy symptoms). Three measurements were taken and the highest measurement recorded on the electronic diary. Daily PNIF is defined as average of PM PNIF and AM PNIF of the next day prior to AM dosing. The Baseline is defined as average of the last 8 readings (4 AM and 4 PM) of PNIF measurement over the four 24-hour periods prior to randomization. Change from Baseline is calculated as the value over the entire treatment period minus the value at Baseline. Analysis was performed using ANCOVA, adjusting for BL value, country, age, and gender.
Time Frame: Baseline (Day 1) and up to 6 weeks
Population: ITT population. Data is presented for the participants available at the time of assessment.
Measure: Least Squares Mean (Standard Error); unit: Liters per minute
Arm/Group | Placebo | Fluticasone Furoate
Number analyzed (Participants) | 150 | 151
Liters per minute | 17.35 (2.13) | 25.72 (2.13)
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Furoate; Test type: Superiority or Other; p = 0.004, ANCOVA; Mean Difference (Final Values) = 8.376, 95% CI 2-sided [2.71 to 14.04]

21. Secondary Outcome: Mean Change From Baseline (Day 1) in AM PNIF Over the Entire Treatment Period
Description: PNIF is the tool for determining the extent of nasal airway obstruction. Participants used a portable hand-held inspiratory flow meter and face mask to measure and record PNIF. AM PNIF measurements was completed and recorded following assessment of allergy symptoms in the AM (prior to taking study medication). Three measurements were taken and the highest measurement recorded on the electronic diary. Baseline AM PNIF is defined as the average of the non-missing values for PNIF during the Baseline period where the Baseline period includes the randomization day and the 3 consecutive days prior to randomization. Change from Baseline is calculated as the value over the entire treatment period minus the value at Baseline. Analysis was performed using ANCOVA, adjusting for Baseline value, country, age, and gender.
Time Frame: Baseline (Day 1) and up to 6 weeks
Population: ITT population. Data is presented for the participants available at the time of assessment.
Measure: Least Squares Mean (Standard Error); unit: Liters per minute
Arm/Group | Placebo | Fluticasone Furoate
Number analyzed (Participants) | 149 | 150
Liters per minute | 16.33 (2.16) | 25.61 (2.17)
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Furoate; Test type: Superiority or Other; p = 0.002, ANCOVA; Mean Difference (Final Values) = 9.280, 95% CI 2-sided [3.52 to 15.04]

22. Secondary Outcome: Mean Change From Baseline (Day 1) in PM PNIF Over the Entire Treatment Period
Description: The PNIF score is the tool for determining the extent of nasal airway obstruction. Participants used a portable hand-held inspiratory flow meter and face mask to measure and record PNIF. PM PNIF measurements was completed and recorded after assessment of allergy symptoms in the PM (12 hours after study medication). Three measurements were taken on each occasion and the highest measurement recorded on the electronic diary. Baseline PM PNIF is defined as the average of the non-missing values for PNIF during the Baseline period where the Baseline period includes the 4 consecutive days prior to randomization. Change from baseline is calculated as the value over the entire treatment period minus the value at Baseline. Analysis was performed using ANCOVA, adjusting for Baseline value, country, age, and gender.
Time Frame: Baseline (Day 1) and up to 6 weeks
Population: ITT population. Data is presented for the participants available at the time of assessment.
Measure: Least Squares Mean (Standard Error); unit: Liters per minute
Arm/Group | Placebo | Fluticasone Furoate
Number analyzed (Participants) | 150 | 147
Liters per minute | 18.51 (2.15) | 26.15 (2.20)
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Furoate; Test type: Superiority or Other; p = 0.009, ANCOVA; Mean Difference (Final Values) = 7.638, 95% CI 2-sided [1.89 to 13.39]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events (nSAEs) were collected from the start of study treatment until follow-up period (Up to 48 days).
Description: SAEs and non-serious AEs were reported for members of the ITT population that comprised of all participants who were randomised to treatment, and received at least one dose of study drug.
Arm/Group | Placebo | Fluticasone Furoate
All-Cause Mortality (participants affected / at risk) | 0/151 | 0/151
Serious Adverse Events (participants affected / at risk) | 0/151 | 1/151
Other Adverse Events (participants affected / at risk) | 66/151 | 77/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=151) | Fluticasone Furoate (N=151)
Acute sinusitis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=151) | Fluticasone Furoate (N=151)
Headache (Nervous system disorders) | 29 | 27
Dizziness (Nervous system disorders) | 1 | 4
Sinus headache (Nervous system disorders) | 2 | 1
Migraine (Nervous system disorders) | 2 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Tension headache (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 13
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Nasal septum ulceration (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 7 | 9
Upper respiratory tract infection (Infections and infestations) | 6 | 3
Influenza (Infections and infestations) | 2 | 3
Viral infection (Infections and infestations) | 1 | 3
Gastroenteritis viral (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 0 | 1
Fungal infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 1 | 0
Nasal candidiasis (Infections and infestations) | 1 | 0
Pharyngeal candidiasis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Purulent discharge (Infections and infestations) | 0 | 1
Rhinovirus infection (Infections and infestations) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 3
Nausea (Gastrointestinal disorders) | 1 | 4
Dyspepsia (Gastrointestinal disorders) | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (General disorders) | 0 | 1
Oral soft tissue disorder (Gastrointestinal disorders) | 1 | 0
Stomach discomfort (Gastrointestinal disorders) | 0 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Pyrexia (General disorders) | 3 | 2
Chest pain (General disorders) | 1 | 1
Fatigue (General disorders) | 0 | 2
Feeling hot (General disorders) | 1 | 1
Thirst (General disorders) | 2 | 0
Chills (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Scab (Skin and subcutaneous tissue disorders) | 1 | 4
Rash (Skin and subcutaneous tissue disorders) | 3 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 3
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 2
Vision blurred (Eye disorders) | 1 | 1
Dry eye (Eye disorders) | 0 | 1
Eye pain (Eye disorders) | 1 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0
Visual disturbance (Eye disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 2
Depression (Psychiatric disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 2
Motion sickness (Ear and labyrinth disorders) | 1 | 0
Food allergy (Immune system disorders) | 0 | 1
Blood pressure increased (Investigations) | 1 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.